CLINICAL TRIAL: NCT05960669
Title: Nerve-sparing, Robot-assisted Radical Prostatectomy Using a Personalized, 3D-printed Prostate Model for Selective Resection of Positive Surgical Margins
Acronym: AURORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AURORA_2018
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
Keywords: prostatectomy; nerve sparing; 3D model; urology; frozen section
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Cohort Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D model guided SR (Experimental): A prostate model was 3D printed from preoperative pelvic MRI data and used during surgery to mark a positive surgical margin and guide secondary resection.
  Interventions: Procedure: 3D model guided secondary resection

INTERVENTIONS:
Procedure: 3D model guided secondary resection — A prostate model was 3D printed from preoperative pelvic MRI data and used during robot-assisted radical prostatectomy to mark a positive surgical margin and guide secondary resection.

SUMMARY:
To optimize precision for secondary resection (SR) in frozen section (FS) controlled nerve-sparing robot-assisted radical prostatectomy (NS-RARP) by using a personalized 3D-printed prostate model.

DETAILED DESCRIPTION:
Background:

Nerve-sparing (NS) robot-assisted radical prostatectomy (RARP) offers optimized oncological and functional outcomes and has become the preferred minimally-invasive approach when available. To maximize oncologic safety in NS-RARP, a frozen section (FS) can be used but does not provide a visual impression of the positive surgical margin (PSM) to guide secondary resection (SR).

Objective:

To optimize precision for secondary resection (SR) in frozen section (FS) controlled nerve-sparing robot-assisted radical prostatectomy (NS-RARP) by using a personalized 3D-printed prostate model.

Design, setting and participants:

100 patients with NS-RARP performed between September 2018 and August 2021 were included in this prospective multicenter cohort study.

Interventions:

A prostate model was 3D printed from preoperative pelvic MRI data and used during surgery to mark a PSM and guide SR.

Outcome Measurements and statistical analysis Endpoints were comparison of the primary surgical margin status in the FS with the tissue of the resulting SR and with the final surgical margin status. Secondary parameters for oncological and erectile outcomes were assessed before and one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* preoperatively planed and intraoperatively performed nerve-sparing approach (at least unilateral)
* suitable pelvic MRI for the creation of a personalized 3D prostate model,
* written patient consent

Exclusion Criteria:

* no nerve sparing performed

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
comparison of the primary surgical margin status in the FS with the tissue of the resulting SR and with the final surgical margin status | 4 weeks

SECONDARY OUTCOMES:
Erectile function | 1 year
  IIEF-5
Oncologic follow-up | 1 year
  PSA Monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Christian CE Engesser, Dr., Principal Investigator — University Hospital, Basel, Switzerland; Jan JE Ebbing, PD Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Universitätsspital Basel Urologie, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No